CLINICAL TRIAL: NCT04590599
Title: A Randomized, Double-blind, Controlled, Parallel-cohort Phase II Clinical Study to Assess the Efficacy and Safety of IBI310 or Placebo Combined With Sintilimab for Advanced Cervical Cancer Subjects Who Have Failed or Cannot Tolerate First-line or Above Platinum-based Chemotherapy
Brief Title: A Phase II Clinical Study to Assess the Efficacy and Safety of IBI310 or Placebo Combined With Sintilimab for Advanced Cervical Cancer Subjects Who Have Failed or Cannot Tolerate First-line or Above Platinum-based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI310E201
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Advanced Cervical Cancer
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI310+Sintilimab (Experimental): IBI310+Sintilimab
  Interventions: Drug: IBI310; Drug: Sintilimab
- Placebo+Sintilimab (Active Comparator): Placebo+Sintilimab
  Interventions: Drug: Placebo; Drug: Sintilimab

INTERVENTIONS:
Drug: IBI310 — IBI310 3 mg/kg,Q3W, for a total of 4 cycles
  Arms: IBI310+Sintilimab
Drug: Placebo — Placebo Q3W, for a total of 4 cycles
  Arms: Placebo+Sintilimab
Drug: Sintilimab — Sintilimab 200mg,Q3W
  Other Names: IBI308

SUMMARY:
This is a randomized, double-blind, controlled, parallel-cohort Phase II clinical study, which is planned to enroll 220 subjects with advanced cervical cancer who have failed or cannot tolerate first-line or above platinum-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the written informed consent form, and can comply with the visits and related procedures specified in the protocol.
2. Aged ≥18 years and ≤75 years.
3. Diagnosed with cervical cancer by histology/cytology.
4. Patients with relapsed or metastatic cervical cancer who have had progressed or relapsed after receiving at least first-line of platinum-based chemotherapy (if a patient has progressed or relapsed during or within 6 months after receiving platinum-based neoadjuvant or adjuvant chemotherapy, she will be deemed to have received first-line treatment).
5. The subject's previous systemic treatment must have ended ≥4 weeks before the first study administration, and the treatment-related AEs have recovered to Common Terminology Criteria for Adverse Events (CTCAE) V5.0 grade ≤1 (except for alopecia and fatigue).

Exclusion Criteria:

1. Diagnosis of other malignant tumors within 5 years before the first administration, excluding radically cured skin basal cell carcinoma, skin squamous cell carcinoma, radically resected carcinoma in situ and/or thyroid papillary carcinoma.
2. Pleural effusion, ascites, and pericardial effusion with clinical symptoms or requiring drainage (patients with effusion that does not require drainage or patients with no significant increase in the effusion within 3 days after stopping drainage can be selected).
3. Patients who are planning to undergo or have previously received organ or bone marrow transplantation.
4. Patients with acute or chronic active hepatitis B or C infection, hepatitis B virus (HBV) DNA> 200 IU/ml or 103 copies/ml; hepatitis C virus (HCV) antibody positive and HCV-RNA level higher than the lower limit of detection. Patients with acute or chronic active hepatitis B or C infection who have received nucleotide antiviral therapy and are below the above standards can be selected.
5. Meningeal metastases or symptomatic central nervous system (CNS) metastases. Patients with asymptomatic brain metastases who do not need treatment with glucocorticoids, anticonvulsants or mannitol after radiotherapy can be enrolled.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Assessed week 6,week 12,week 18 ,and every 9 weeks (or every 12 weeks after 54 weeks of treatment) for duration of study participation which is estimated to be 24 months.
  Objective response rate (ORR) assessed by the Independent Radiological Review Committee (IRRC) according to the Response Evaluation Criteria in Solid Tumors (RECIST) V1.1
Objective response rate (ORR) | Assessed week 6,week 12,week 18 ,and every 9 weeks (or every 12 weeks after 54 weeks of treatment) for duration of study participation which is estimated to be 24 months.
  ORR assessed by the investigator according to the RECIST V1.1

SECONDARY OUTCOMES:
Disease Control Rate（DCR） | Assessed week 6,week 12,week 18 ,and every 9 weeks (or every 12 weeks after 54 weeks of treatment) for duration of study participation which is estimated to be 24 months.
  DCR assessed by the investigator and IRRC according to the RECIST V1.1

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Innovent Biologics, Inc., Suzhou, Jiangsu
  - Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital）, Zhenjiang

REFERENCES:
- [Derived] Li H, Xu Y, Jiao X, Xu Q, Peng Z, Tang Y, Zhang J, Huang B, Shen Y, Chang B, Xia B, Duan W, Wang D, Zhu L, An R, Zhang G, Tang Y, Huang J, Qiu H, Wang L, Huang Y, Li G, Qian J, Sun L, Zheng H, Lou G, Zhang Y, Chen Y, Lu L, Cheng Y, Liu J, Zhao W, Ji J, He A, Wang K, Yu G, Zhu H, Ma C, Yuan J, Wang X, Zhang H, Ma X, Cai C, Yin K, Xie H, Wang Y, Wang S, Li L, Zhou H, Wang J, Zhu J, Ma D, Gao Q. IBI310 plus sintilimab vs. placebo plus sintilimab in recurrent/metastatic cervical cancer: A double-blind, randomized controlled trial. Med. 2025 May 9;6(5):100573. doi: 10.1016/j.medj.2024.100573. Epub 2025 Jan 18. PMID 39827881